CLINICAL TRIAL: NCT02356120
Title: The Inter-observer Reliability and Diagnostic Accuracy of Tricuspid Annular Plane Systolic Excursion in Patients With Suspected Pulmonary Embolus in the Emergency Department
Brief Title: Inter-Observer Reliability and Accuracy of Tricuspid Annular Plane Systolic Excursion in Patients With Suspected PE in the ED
Status: Withdrawn | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1412015010
Record Dates: First submitted 2015-01-30; First posted 2015-02-05 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected Pulmonary Embolus: Patients with suspected pulmonary embolus who are getting a CTPA
  Interventions: Other: Echocardiogram

INTERVENTIONS:
Other: Echocardiogram — Tricuspid annular plane systolic excursion will by measured by emergency physician performed echocardiogram

SUMMARY:
The purpose of this study will be to evaluate the measurement of tricuspid annular plane systolic excursion (TAPSE) by emergency physician performed echocardiogram on patients with suspected pulmonary embolism (PE) who are scheduled to get a computed tomography of the pulmonary arteries (CTPA)

DETAILED DESCRIPTION:
This will be a prospective observational cohort study aimed at determining the utility and reproducibility of TAPSE, in patients who present to the emergency department with suspected pulmonary embolism (PE). The gold standard diagnostic test for PE is computed tomography of the pulmonary arteries (CTPA). Any patient for whom a CTPA is ordered because of suspected PE is eligible for study inclusion

ELIGIBILITY:
Inclusion Criteria:

* Concern for PE by attending physician and CTPA ordered

Exclusion Criteria:

* If patient is under the age of 18, a prisoner, or a ward of the state
* CTPA ordered but not performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population will consist of a convenience sample, taken when study investigators are available, of all those patients for whom suspicion of PE is high enough that their attending physician has ordered a CTPA in the ED
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of TAPSE (The association of TAPSE measurements with a diagnosis of PE will be explored using multivariate analysis) | 0 days
  The association of TAPSE measurements with a diagnosis of PE will be explored using multivariate analysis

SECONDARY OUTCOMES:
Inter-Observer Agreement (To assess the interobserver reproducibility of measuring TAPSE, intra-class correlation coefficients and Bland-Altman analysis will be performed.) | 0 days
  To assess the interobserver reproducibility of measuring TAPSE, intra-class correlation coefficients and Bland-Altman analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Moore, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States